CLINICAL TRIAL: NCT06176651
Title: Evaluation of Miebo (Perfluorohexyloctane) Eyedrops in Habitual Contact Lens Wearers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gordon Schanzlin New Vision (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSNVI-MIEBO1
Record Dates: First submitted 2023-12-08; First posted 2023-12-20 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye; Dry Eye, Evaporative; Dry Eye Disease; Evaporative Dry Eye; Evaporative Dry Eye Disease; Kerato Conjunctivitis Sicca
Keywords: Contact Lens; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — perfluorohexyl-octan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Arm (Experimental): This is a single arm open label study with no randomization or control group. All participants will receive the Miebo eye drop for use while enrolled in the study.
  Interventions: Drug: Miebo

INTERVENTIONS:
Drug: Miebo — Subjects will be instructed to use the Miebo eye drop four times per day in both eyes during their participation in clinical trial. The subjects will be required to remove their contact lenses prior to instillation of the Miebo eye drop and must wait 30 minutes before reinserting their contact lenses.

SUMMARY:
Miebo (Perfluorohexyloctane) is a novel, non-aqueous, single entity, preservative free, ophthalmic drop. This drop was recently approved by the Food and Drug Administration (FDA) for the treatment of Meibomian Gland Disease (MGD).

All published data on Miebo has been done in non-contact lens wearers. As contact lens dropout rates seem to be an ongoing problem for practitioners, we are performing this study utilizing this novel new drug with contact lens patients to determine if the drops assist comfort in typical soft contact lens wearing patients. If the study determines that Miebo assists in the overall comfort of contact lens patients this could be a possible way to help keep patients in their contact lenses longer.

DETAILED DESCRIPTION:
The study design is a single center, open label, double arm study with no control and no randomization. We will enroll 50 patients who are adjusted contact lens wearers who have corrected visual acuity of 20/25 or better at distance. 25 patients will be in daily disposable contact lens of varied manufacturers. The other 25 will be in monthly disposable contact lenses of varied manufacturers. Subjects will insert the Miebo eye drops four times a day, and with their contact lenses removed every day. Subjects will be required to wait at least 30 minutes before inserting their lenses after drop use. Subjects will be seen on day 0 for initial screening, on day 7 and finally on day 30. The window for visits on day 7 is +/-3 and for day 30 +/- 7 days. Visits on day 7 and 30 will be conducted at least one hour post Miebo insertion. Overall vision and comfort will be assessed during the study. The primary endpoint is to show that Miebo eye drops are safe to use in contact lens wearers. The secondary endpoint is to show changes in comfort in contact lens wearing individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years of age
* Habitual contact lens wear for ≥ 60 days
* Willing to sign the informed consent form and is deemed capable of complying with the requirements of the study protocol.

Exclusion Criteria:

* Previous use or known allergy to Miebo
* Subjects with corneal abnormality or eye pathology that would affect the outcome in the investigator's opinion.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this clinical trial is to evaluate the safety of Miebo for contact lens wearers. | 30 days
  This assessment will be conducted by comparing the total corneal fluorescein staining (tCFS) score for each participant before the initiation of Miebo usage and after one month of consistent use. The total corneal fluorescein staining (tCFS) score will allow quantitative assessment of the extent of damage or irregularities on the corneal surface if present. Safe use of Miebo will be determined by an increase of tCFS score for each eye of 10% or less compared to the baseline tCFS score.

SECONDARY OUTCOMES:
The secondary outcome of this clinical trial is to evaluate the tolerability of Miebo for contact lens wearers. | 30 days
  This assessment will be conducted by comparing the results of the CLDEQ-8 (Contact Lens Dry Eye Questionnaire-8) for each participant before the initiation of Miebo usage and after one month of consistent use. The Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) is a standardized and validated questionnaire designed to assess the impact of dry eye symptoms specifically in individuals who wear contact lenses. This questionnaire serves as a valuable tool to quantify and understand the subjective experiences of contact lens wearers in relation to dry eye symptoms. Successful tolerability will be quantified by am increase in the total CLDEQ-8 score of 10% or less compared to the baseline CLDEQ-8 score.

CONTACTS AND LOCATIONS:
Locations (1):
- Gordon Schanzlin New Vision Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No